CLINICAL TRIAL: NCT01758250
Title: Mechanistic Study: Non-Invasive Cutaneous Microvascular and Fibrosis Imaging of Patients With Systemic Sclerosis, Sickle Cell Disease and Chronic Graft-Versus-Host Disease (GVHD) Compared to Healthy Subjects
Brief Title: Microvascular and Fibrosis Imaging Study
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00039256
Record Dates: First submitted 2012-12-26; First posted 2013-01-01 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-05

CONDITIONS: Autoimmune Diseases; Sickle Cell Disease; Chronic Graft Versus Host Disease
Keywords: Autoimmune diseases with cutaneous involvement; Systemic sclerosis; Scleroderma; Morphea; Dermatomyositis; Cutaneous lupus; Vasculitis; Sickle Cell Disease; Graft versus Host Disease
MeSH Terms: conditions — Autoimmune Diseases; Anemia, Sickle Cell; Bronchiolitis Obliterans Syndrome; Scleroderma, Systemic; Scleroderma, Diffuse; Scleroderma, Localized; Dermatomyositis; Vasculitis; Graft vs Host Disease | interventions — Laser-Doppler Flowmetry; Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Systemic Sclerosis: Patients with SSc will have imaging studies performed at baseline and at 3, 6, 9, 12, 15, 18, 21 and 24 months.
  Interventions: Other: Acoustic Radiation Force Impulse (ARFI); Other: Laser Doppler Flowmetry (LDF); Other: Laser Doppler Perfusion Imaging (LDI); Other: Optical Coherence Tomography (OCT); Other: Orthogonal Polarization Spectral Imaging (OPSI); Other: Nail fold video capillaroscopy (NVC)
- GVHD: Patients with GVHD will have imaging studies performed at baseline and at 3, 6, 9, 12, 18 and 24 months.
  Interventions: Other: Acoustic Radiation Force Impulse (ARFI); Other: Laser Doppler Flowmetry (LDF); Other: Laser Doppler Perfusion Imaging (LDI); Other: Optical Coherence Tomography (OCT); Other: Orthogonal Polarization Spectral Imaging (OPSI); Other: Nail fold video capillaroscopy (NVC)
- Undergoing HSCT: Patients who are about to undergo HSCT will have imaging studies performed at 1 week pre-transplantation, day 40 and 80 post transplantation and at 3 months, 6 months, 12 months 18 months and 24 months post-transplant.
  Interventions: Other: Acoustic Radiation Force Impulse (ARFI); Other: Laser Doppler Flowmetry (LDF); Other: Laser Doppler Perfusion Imaging (LDI); Other: Optical Coherence Tomography (OCT); Other: Orthogonal Polarization Spectral Imaging (OPSI); Other: Nail fold video capillaroscopy (NVC)
- Controls: Healthy Controls and Controls with hematologic and solid organ malignancies and dermatitis will have imaging studies performed at a single point in time.
  Interventions: Other: Acoustic Radiation Force Impulse (ARFI); Other: Laser Doppler Flowmetry (LDF); Other: Laser Doppler Perfusion Imaging (LDI); Other: Optical Coherence Tomography (OCT); Other: Orthogonal Polarization Spectral Imaging (OPSI); Other: Nail fold video capillaroscopy (NVC)
- Sickle cell disease: Patients with SCD will have imaging studies performed at baseline and at 3, 6, 9, 12, 15, 18, 21 and 24 months.
  Interventions: Other: Acoustic Radiation Force Impulse (ARFI); Other: Laser Doppler Flowmetry (LDF); Other: Laser Doppler Perfusion Imaging (LDI); Other: Optical Coherence Tomography (OCT); Other: Orthogonal Polarization Spectral Imaging (OPSI); Other: Nail fold video capillaroscopy (NVC)
- Cutaneous fibrosing disorder: Patients with active cutaneous fibrosing disorder will have imaging studies performed at a single point in time.
  Interventions: Other: Acoustic Radiation Force Impulse (ARFI); Other: Laser Doppler Flowmetry (LDF); Other: Laser Doppler Perfusion Imaging (LDI); Other: Optical Coherence Tomography (OCT); Other: Orthogonal Polarization Spectral Imaging (OPSI); Other: Nail fold video capillaroscopy (NVC)

INTERVENTIONS:
Other: Acoustic Radiation Force Impulse (ARFI)
Other: Laser Doppler Flowmetry (LDF)
Other: Laser Doppler Perfusion Imaging (LDI)
Other: Optical Coherence Tomography (OCT)
Other: Orthogonal Polarization Spectral Imaging (OPSI)
Other: Nail fold video capillaroscopy (NVC)

SUMMARY:
In this study, Laser Doppler Flowmetry (LDF), Laser Doppler Imaging (LDI), Orthogonal Polarization Spectral Imaging (OPSI), Nail fold video capillaroscopy (NVC) and Optical Coherence Tomography (OCT) will be used to assess differences in microvascular function and density of oral mucosa and skin in subjects with 1) autoimmune diseases with cutaneous involvement: systemic sclerosis (SSc), morphea, dermatomyositis, cutaneous lupus and vasculitis, 2) sickle cell disease (SCD) and 3) chronic graft-versus-host disease (GVHD) compared to healthy subjects. The microvascular changes will be compared to overall treatment response in patients with scleroderma and chronic GVHD as assessments will be made before and after the patients start treatment for their diseases and determine if these imaging techniques provide valuable and reproducible data when assessing a patient's response to treatment for those diseases. In addition, the application of Acoustic Radiation Force Impulse (ARFI) in determining cutaneous thickness in patients with SSc, GVHD and morphea will be evaluated.

The investigators hypothesize that the vascular and dermal structures are altered in patients with autoimmune disease, SCD and chronic GVHD. In addition, they hypothesize that imaging modalities such as LDF, LDI, OCT, NVC, OPSI and ARFI can quantify such structural alterations and can be used to 1) detect early disease activity, 2) quantify and assess response to therapy and 3) quantify and correlate with overall disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects above the age of 18 who are capable of giving informed consent with one of the following conditions: Scleroderma, Graft vs Host Disease, Sickle Cell Disease, Morphea, Connective Tissue Disease with cutaneous manifestations: cutaneous lupus, dermatomyositis, vasculitis, patients who are undergoing HSCT, or patients with a diagnosis of hematologic and non-hematologic malignancies without GVHD
* Control patients include normal healthy controls above the age of 18 who are capable of giving informed consent.

Exclusion Criteria:

* Patients who experience discomfort, will be prone to experience discomfort or cannot tolerate the position required for the imaging studies.
* Subjects unable to provide informed consent.
* Smokers, patients unable to tolerate caffeine avoidance for the day of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient population at Duke University Medical Center and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Microvascular density in oral mucosa and skin | over 24 months
  Microvascular density as evaluated using LDF, LDI, OPSI, OCT, NVC and AFRI, will be compared between subjects with and without disease.
Microvascular Perfusion in oral mucosa and skin | over 24 months
  Microvascular perfusion as evaluated using LDF, LDI, OPSI, OCT, NVC, and AFRI, will be compared between subjects with and without disease.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Sullivan, MD, Principal Investigator — Duke University; Adela Cardones, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States